CLINICAL TRIAL: NCT01324635
Title: Phase I, Dose Finding Trial of the Combination of Panobinostat and Stereotactic Radiation in the Treatment of Brain Tumors
Brief Title: Panobinostat and Stereotactic Radiation Therapy in Treating Patients With Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Arm A - reached goal; Arm B - poor accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11D.100; 2010-38 (Other: CCRRC); JT 2158 (Other: JeffTrial Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-29 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Glioma; High-grade Meningioma; Brain Metastasis
Keywords: glioma; meningioma; brain metastasis; stereotactic; radiotherapy; radiosurgery
MeSH Terms: conditions — Glioma; Brain Neoplasms; Meningioma | interventions — Panobinostat; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (panobinostat, multiple fractions of SBRT) (Experimental): Patients receive panobinostat PO thrice weekly for 2 weeks and undergo 10 fractions of SBRT over 2 weeks (recurrent gliomas) OR 30 fractions of SBRT over 6 weeks (high grade meningiomas).
  Interventions: Drug: Panobinostat; Radiation: Stereotactic body radiation therapy; Procedure: Quality-of-life assessment
- Arm B (panobinostat, stereotactic radiosurgery) (Experimental): Patients receive panobinostat as in Arm A and undergo a single fraction of stereotactic radiosurgery on day 1 of week 1.
  Interventions: Drug: Panobinostat; Procedure: Quality-of-life assessment; Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Drug: Panobinostat — Given PO
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Radiation: Stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
  Arms: Arm A (panobinostat, multiple fractions of SBRT)
Procedure: Quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Radiation: Stereotactic radiosurgery — Undergo stereotactic radiosurgery
  Arms: Arm B (panobinostat, stereotactic radiosurgery)

SUMMARY:
This is an open label phase I clinical trial with two arms, representing single and fractionated radiation therapy (Figure 4.1). Within each arm the radiation dose is pre-determined and not escalated. Panobinostat will be administered orally 3 times a week for 2 weeks. Panobinostat will be dose-escalated independently in each arm. There is no intra-patient dose escalation.

Recurrent gliomas (Arm A) will be treated according to the Jefferson protocol for re-irradiation, 10 fractions each of 3.5Gy delivered over 2 weeks. Panobinostat will be administered orally three times a week for 2 weeks, starting on day 1 or 2 of radiation therapy. High-grade meningiomas (Arm A) will be treated with 6 weeks/30 fractions of fractionated radiation therapy, to a total dose of between 54 Gy and 60 Gy in fractions of either 1.8Gy or 2Gy. Panobinostat will be administered orally three times a week for 2 weeks, starting on the day of 1st fraction of radiation.

Large brain metastases (Arm B) will be treated with a single fraction of radiosurgery. Panobinostat will be administered orally three times a week for 2 weeks, starting on the day of radiation. The radiosurgery may be delivered by either LINAC, gamma-knife, cyber-knife or tomotherapy technology.

DETAILED DESCRIPTION:
Brain tumors, both primary and metastatic present a therapeutic challenge. Radiation therapy plays a major role in management of both entities. Nonetheless, local control remains sub-optimal in a large proportion of patients. Over the previous decade there has been a great deal of progress regarding 1) precision in the localization and targeting of brain lesions with radiation, 2) increased use of single/hypofractionation schedules and 3) combining fractionated conformal radiation with targeted agents. This trial utilizes a novel approach - the combination of an HDAC inhibitor (Panobinostat) with stereotactic radiosurgery. The combination blends the advantages of extreme high precision radiation with a potent targeted agent - promising enhanced efficacy with minimal toxicity. The investigators will examine the combination in three settings, in all of which current standard of care is sub-optimal:

1. Recurrent glioma
2. High grade meningioma
3. Large brain metastases from solid malignancies

Histone deacetylase (HDAC) inhibitors, including Panobinostat, radiosensitize tumor cells both in vitro and in vivo. HDAC inhibitors modify the expression of approximately 8% of the transcriptome83. In particular, they have been shown to down regulate expression of the DNA repair enzyme rad51, possibly explaining their radiosensitization properties. It is thought that Panobinostat radiosensitizes through an epigenetic mechanism. Since the target of HDAC inhibitors includes many proteins beyond histones, many prefer the name "deacetylase inhibitors", (DAC).

There are several lines of evidence suggesting HDAC inhibitors cross the BBB. The anticonvulsant valproic acid, a member of the short chain fatty acid class of HDAC inhibitors, has a well-recognized capacity to cross the BBB. HDAC inhibitors are also being studied in Huntington's disease. Panobinostat is able to cross the blood-brain-barrier and influence gene expression in rodents.

When combining radiation therapy with systemic agents it is generally considered important that there is a high concentration of drug present at, or just before, the time of irradiation. The goal is to use panobinostat as a radiosensitizer, not a single systemic agent. The investigators will administer oral panobinostat 3 times weekly for 2 weeks. This is an open label phase I clinical trial with two arms, representing single and fractionated radiation therapy (Figure 4.1). Within each arm the radiation dose is pre-determined and not escalated. Panobinostat will be administered orally 3 times a week for 2 weeks. Panobinostat will be dose-escalated independently in each arm. There is no intra-patient dose escalation.

Recurrent gliomas (Arm A) will be treated according to the Jefferson protocol for re-irradiation, 10 fractions each of 3.5Gy delivered over 2 weeks. Panobinostat will be administered orally three times a week for 2 weeks, starting on the day of 1st fraction of radiation. High-grade meningiomas (Arm A) will be treated with 6 weeks/30 fractions of fractionated radiation therapy, to a total dose of between 54 Gy and 60 Gy in fractions of either 1.8Gy or 2Gy. Panobinostat will be administered orally three times a week for 2 weeks, starting on the day of 1st fraction of radiation.

Large brain metastases (Arm B) will be treated with a single fraction of radiosurgery. Panobinostat will be administered orally three times a week for 2 weeks, starting on the day of radiation. The radiosurgery may be delivered by either LINAC, gamma-knife, cyber-knife or tomotherapy technology.

Radiation treatment: definition of target volumes:

Recurrent gliomas (Arm A) If progression is diagnosed with the development of new enhancing tumor: The gross tumor volume (GTV) will be defined by the new contrast-enhanced T1 abnormality on the post-operative MRI scan. This will generally include the surgical cavity margins from the most recent surgical procedure. If progression is diagnosed with the development of new non-enhancing tumor: volumes will be defined through careful comparison of new and previous MRI scans in consultation with a neuro-radiologist. This will generally include the surgical cavity margins from the most recent surgical procedure.

The GTV will then be expanded by an additional margin of 5.0 mm to create the PTV. This 5mm margin may be reduced, or eliminated around natural barriers to tumor growth such as the skull, ventricles, falx, etc, and also to allow sparing of the optic nerve/chiasm or other critical structure at the discretion of the treating physician. The minimum dose to the PTV will be 95% of the prescription dose (35Gy). The maximum dose to the PTV will be 110%. Any beam arrangement and set of energies that accomplishes these criteria is allowed.

High-grade meningiomas (Arm A) Target volumes will be based upon postoperative-enhanced MRI (unless only biopsy was performed). Preoperative imaging may be used for correlation and improved identification. The gross tumor volume (GTV) will be defined by the tumor bed on the postoperative- enhanced MRI and is to include any residual nodular enhancement. Cerebral edema is not to be specifically included within the GTV. The "dural tail" may or may-not be included depending on physician preference. The clinical target volume (CTV) will be the GTV plus a margin of between 1.0 cm and 2.0cm according to physician preference. The CTV margin may be reduced to 0.5 cm around natural barriers to tumor growth such as the skull. The planning target volume (PTV) is an additional margin of 3.0 to 5.0 mm, depending upon localization method and reproducibility. PTV margins account for variations in set-up and reproducibility. The CTV/PTV margins way be modified to allow sparing of the optic nerve/chiasm or other critical structure at the discretion of the treating physician.

The minimum dose to the PTV will be 95% of the prescription dose (35Gy). The maximum dose to the PTV will be 110%. Any beam arrangement and set of energies that accomplishes these criteria is allowed.

Large brain metastases (Arm B) Single fraction radiosurgery doses will be in accordance with prescriptions from RTOG radiosurgery trial 90-058. Metastases larger than 2 cm but equal to or smaller than 3 cm will be treated with 18•0 Gy; and metastases larger than 3 cm and less than or equal to 4 cm will be treated to a prescription dose of 15.0 Gy. Radiation therapy should be planed in accordance with standard radio-surgical principals, i.e. prescribed to the 50% isodose line for gamma-knife and 90% isosurface for LINAC based systems.

6.3 Technical aspects of radiation therapy Fractionated treatment will be highly conformal external beam radiation therapy (EBRT) delivered with either gamma-knife, tomotherapy, cyberknife or megavoltage LINAC radiation therapy machines of energy ≥ 6 MV. Any standard technique of dose planning including conformal dynamic arcs, 3D-CRT or IMRT may be used.

For single fraction treatments cyber-knife, LINAC, tomotherapy or gamma-knife based radiosurgery may be used.

Normal tissue constraints Arm A, Recurrent glioma The brain stem: no more than 1cm3 should receive more than 30Gy; optic chiasm and optic nerves should not receive more than 25Gy, unless included in the target volume.

Arm A, High-grade meningioma Lenses 7Gy, Retinae 50Gy, Optic Nerves 55Gy, Optic Chiasm 56Gy, Brainstem 60Gy Arm B, Single fraction Brain stem no more than 1cm3 should receive more than 10Gy; optic chiasm and optic nerves no more than 8 Gy;

In the event that an organ at risk (OAR) is in immediate proximity to a PTV such that dose to the OAR cannot be constrained within protocol limits, the final decision is left to the treating physician to weigh up potential treatment toxicity versus under-coverage of target volume.

Panobinostat for oral administration will be provided by Novartis. Medication labels will comply with US legal requirements and be printed in English. They will supply no information about the patient. The storage conditions for study drug will be described on the medication label, and the investigator's brochure, edition #5 19-Jun-2009.

Panobinostat should be administrated after at least 2-hour fast, and subjects will continue the fast for 2 more hours. If the patient misses one or more doses of panobinostat and it is before the next dose of panobinostat is due, the patient should take the make up dose at the earliest time, then resume the protocol schedule. If patient misses one or more doses of panobinostat, and the patient is due for the next dose of panobinostat, the patient should resume the protocol schedule without making up for the missing dose/doses. If the patient misses one or more panobinostat doses and it is past the scheduled last dosing time of the panobinostat, the patient should stop panobinostat without making up for the missing dose/doses.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is > or = 18 years
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of < or = 2
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
4. Patients must meet the following laboratory criteria:

   * Hematology:

     * Neutrophil count of > 1500/mm3
     * Platelet count of > 100,000/mm3L
     * Hemoglobin > or = 9 g/dL
   * Biochemistry:

     * AST/SGOT and ALT/SGPT < or = 2.5 x upper limit of normal (ULN) or < or = 5.0 x ULN if the transaminase elevation is due to disease involvement
   * Serum bilirubin < or = 1.5 x ULN
   * Serum creatinine < or = 1.5 x ULN or 24-hour creatinine clearance > or = 50 ml/min
   * Total serum calcium (corrected for serum albumin) or ionized calcium > or = LLN
   * Serum potassium > or = LLN
   * Serum sodium > or = LLN
   * Serum albumin > or = LLN or 3g/dl
   * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
5. Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment. and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
7. Pathologic diagnosis and other conditions relating to the different arms of the study:

   * Arm A Recurrent glioma: Pathological diagnosis of glioma (grade 2-4) is required. All patients are required to have initially undergone fractionated radiation therapy, to between 55 Gy to 70 Gy in fractions of 1.8-2 Gy as part of 'first line therapy'. The diagnosis of 'recurrence' is to be made by the treating physician on the basis of radiological and clinical data. Measurable disease is not required.
   * Arm A High-grade meningioma: Pathological diagnosis of high-grade meningioma, as defined by WHO grade 2 or 3 (also known as atypical and anaplastic/malignant meningioma). WHO grade 1 meningiomas with an elevated Ki67 proliferation rate of > or = 8% are also considered high-grade for the purposes of this trial, due to their poor prognosis32, 86-88. The meningioma may be treated in the scenario of either adjuvant treatment (radiation therapy following complete / sub-total / biopsy only resection) or recurrent disease (re-growth following surgery alone). Measurable disease is not required.
   * Arm B Large brain metastases: Pathological diagnosis of malignancy is required, from either the primary tumor or a metastasis. A radiological diagnosis (CT or MRI scan) of one of more brain metastases is required. At least one of the brain metastases to be treated as part of this study must be 2.5cm or larger in maximal diameter. The brain metastasis/es to be treated may not be more than 4cm in maximal diameter, as assessed by CT or MRI scan. The brain metastasis may either be un-resected or partially resected, provided that the target lesion (which may include a resection cavity) remains between 2.5 and 4cm in diameter, as defined in section 6. Whole brain radiation therapy may or may-not have been delivered prior to entering this protocol.

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
3. Impaired cardiac function including any one of the following:

   * History or presence of sustained ventricular tachyarrhythmia.
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as HR < 50 bpm. Patients with pacemakers are eligible if HR > or = 50 bpm.
   * Screening ECG with a QTc > 450 msec
   * Right bundle branch block + left anterior hemiblock (bifascicular block)
   * Patients with myocardial infarction or unstable angina < or = 6 months prior to starting study drug
   * Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
4. Uncontrolled hypertension
5. Concomitant use of drugs with a risk of causing torsades de pointes
6. Patients with unresolved diarrhea > or = grade 2
7. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
8. Other concurrent severe and/or uncontrolled medical conditions
9. Patients who have received chemotherapy, any investigational drug or undergone major surgery < 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
10. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral panobinostat.
11. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
12. Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
13. Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
14. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
15. Allergy to MRI contrast agent.
16. Any anti-cancer treatment within 2 weeks of initiating treatment as part of this trial, including cytotoxic chemotherapy (e.g. temozolomide), radiation therapy (single fraction or fractionated), and biological therapies (e.g. mono-clonal antibodies, tyrosine kinase inhibitors, interferon). Hormonal therapies (e.g. in breast and prostate cancer) are allowed both prior to and during treatment.
17. Exclusion criteria specific to arms of the trial:

    * Arm A Recurrent glioma: The subject has received more than one prior course of radiation therapy within the target volume to be treated as part of this protocol. Additional courses of radiation therapy (single fraction or fractionated) are permitted if outside of the volume to be treated.
    * Arm A High-grade meningioma: The subject has received a prior course of radiation therapy within the target volume to be treated as part of this protocol.
    * Arm B Large brain metastases: The subject has received a prior course of radiation therapy within the target volume to be treated as part of this protocol, aside from whole brain radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated does (MTD) of panobinostat, defined as one level below at which 2 of 6 patients experience a dose-limiting toxicity (DLT) | Up to 30 days after the completion of study treatment
  Assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Dose-limiting toxicities as defined by the NCI CTCAE version 4.0 | Up to 30 days after the completion of study treatment
Overall survival | Assessed up to 2 years
  Analyzed using Kaplan-Meier estimates
Progression free survival (PFS) | Assessed up to 2 years
  Analyzed using Kaplan-Meier estimates
Response as defined by RECIST criteria | 8 weeks after completion of study treatment
  A 2-sided exact 95% confidence interval will be computed.
Response as defined by RECIST criteria | Assessed up to 2 years
  A 2-sided exact 95% confidence interval will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org